CLINICAL TRIAL: NCT04336566
Title: Renal Function in Chronic Kidney Disease and the Effect of Exogenous Melatonin Administration (REM TRIAL)
Brief Title: Renal Effects of Melatonin Trial in Chronic Kidney Disease
Acronym: REM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10584
Record Dates: First submitted 2020-03-16; First posted 2020-04-07 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, data manager/monitor, principle investigator all blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): 5mg dose of melatonin manufactured by Good Neighbor Pharmacy
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Good Neighbor Pharmacy placebo tablet that looks the same without active ingredient
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin 5mg
  Arms: Melatonin
Dietary Supplement: Placebo — Comparable Good Neighbor Pharmacy placebo tablet
  Arms: Placebo

SUMMARY:
This will be a prospective, double blinded, randomized, controlled pilot study to determine if there is any correlation between melatonin administration and proteinuria.

DETAILED DESCRIPTION:
Investigators plan to enroll up to 100 eligible participants in this pilot trial with 50 participants randomized to receive melatonin and 50 patients randomized to receive a placebo. Participants will be randomized on a rolling basis; meaning, once participants agree to enroll in the study, the participant will be placed randomly into either group.

ELIGIBILITY:
Inclusion Criteria:

* Are between ages 18 and up with chronic kidney disease (CKD) I-III (stage 3 kidney disease, kidney dysfunction)
* Random urine microalbumin of 30 mcg or greater (protein in the urine)
* Have ability to complete a sleep survey
* Currently not on melatonin therapy.

Exclusion Criteria:

* End Stage Renal Disease
* CKD Stage IV (stage 4 with severe kidney dysfunction)
* Severe liver disease
* Chronic dialysis therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Change in Albuminuria | 6 months
  protein in urine

SECONDARY OUTCOMES:
Surveys including Pittsburgh Sleep Quality Index (PSQI) questionnaire | 6 months
  Scale 0-21, higher scores indicate worse sleep quality
Sodium levels | 6 months
  electrolyte in blood
Urinalysis | 6 months
  To asses electrolyte and protein levels
Creatinine levels | 6 months
  serum blood
Blood Urea Nitrogen (BUN) levels | 6 months
  Blood Urea Nitrogen
Potassium levels | 6 months
  mineral in blood
Bicarbonate levels | 6 months
  base found in blood
Chloride levels | 6 months
  electrolyte in blood

CONTACTS AND LOCATIONS:
Overall Officials: Krishna M Baradhi, MD, Principal Investigator — OUHSC
Locations (1):
- University of Oklahoma School of Community Medicine, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No